CLINICAL TRIAL: NCT03065439
Title: The Association Between STarT Back Tool Subgroups of Patients With Low Back Pain and Postural Stability Under Conditions of Sensory Deprivation and Cognitive Load
Brief Title: The Association Between STarT Back Tool Subgroups and Postural Stability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Principal Investigator, Allan Riis, Post doc, Aalborg University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: AllanRiis_6
Record Dates: First submitted 2017-02-17; First posted 2017-02-28 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Low Back Pain, Postural
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: This is a double blinded experimental study comparing sub-groups of patients with low back pain
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Balance testing will be performed and data saved without the testers knowing the results. Afterwards the testers will ask patients to fill in questionnaires. An assessor (not participating in testing) will be cleaning the data and establishing the models without knowledge of the SBT score. The STarT Back score will be cleaned, saved in another data set and established by another assessor. When agreed upon the model, the two data sets will be merged.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STarT Back Tool group 3 (Experimental): Patients scored as high risk patients by the STarT Back Tool
  Interventions: Diagnostic Test: Static balance testing
- STarT Back Tool groups 1+2 (Experimental): Patients scored as low risk or medium risk patients by the STarT Back Tool
  Interventions: Diagnostic Test: Static balance testing

INTERVENTIONS:
Diagnostic Test: Static balance testing — Postural sway will be measured using a force plate (Metitur Good Balance System®).

SUMMARY:
Purpose This trial study the association between SBT subgroups and postural stability. It is theorized that cognitive impairment is more pronounced among patients in SBT group three compared to SBT group one and two. Therefore, it is hypothesized that challenging patients' balance will have a greater impact on the postural sway among patients in SBT group three compared to SBT group one and two in conditions where sensory information is reduced and cognitive load is increased.

DETAILED DESCRIPTION:
Globally low back pain (LBP) and neck pain are the leading causes of disability (1). Consequently, improvements in the assessment and treatment of LBP can have an extensive impact. Patients with LBP constitute a heterogeneous group and to improve treatment there is much focus on identifying subgroups of patients and tailor treatment accordingly. An example of this is the STarT Back Tool (SBT) which has been translated to more than 20 languages and is probably the most used tool for subgrouping of patients with LBP. The SBT sub-groups patients into three groups with a progressing need for treatment. Patients in group one should be given information on LBP and advice to stay active, patients in group two are also recommended supplementary treatment in primary care, and in addition patients in group three need attention to psycho-social issues (2-3). Accordingly to the SBT, patient in group three should be treated with cognitive therapy by a physiotherapist undergoing special training. This training includes mentorship and professional support to enable physiotherapists to elicit and address complex issues in patients with psycho-social barriers to recovery. Subgrouping by SBT and thereby treating patients in group three with cognitive therapy has been found effective in improving their functional outcomes (4-5).

Patients with LBP have found to have different postural control strategies than patients without LBP especially during tasks involving increased task complexity (6-7). However, some studies have not found decreased postural control among patients whit LBP (8-9). Heterogeneous study populations may explain the discrepancy in findings especially if subgroups of patients with LBP have affected postural control while other subgroups are not affected.

Patients with pain often present with some degree of cognitive impairments which could limit the extent to which daily activities could be performed. This may be particularly present among SBT group three patients. Cognitive impairments have been associated with decreased function and consequently reduced balance in elderly, indicating that postural stability requires significant amount of cognitive resource. Since the cognitive resources are limited, if additional tasks compete for these resources, performance in one or more tasks can become affected. The conscious interpretation of (or attention towards) painful stimulations is a costly process that uses significant amount of the cognitive resources available which could impair physical performance. Consequently, this may lead to additional postural sway and thereby restricted balance.

After given written informed consent patients fill in a questionnaire including age, gender, educational level (bachelor, yes/no), employment, sick leave, co-morbidity (other than LBP, yes/no), pain duration (2-6 weeks/sub-acute or chronic), pain intensity (NPR), Roland Morris Disability Questionnaire (23 question, RMDQ), self-reported health status (EQ-5D visual analogue scale). After filling in the questionnaire patients will be asked to take of their jacket and shoes and to empty their pockets, before measuring height, weight, and testing for static balance.

Postural sway will be measured using a force plate (Metitur Good Balance System®). The force plate will be placed with a distance of 100 cm to a wall in front of the patient and with more than 100 cm of free space to the sides and behind the force plate. The force plate, an equilateral triangle (800 mm), had four strain gauge transducer signals converted by a three-channel DC amplifier and transformed to digital data (50 Hz) and subsequently filtered digitally, using a three-point median filter and IRR filter, with 20 Hz cut-off frequency. On the wall in front of the patient a 12 cm circular green plate will be place in the patients' eye level. Patients will be asked to stand with their feet as closed positioned as possible, without lifting their feet, and to focus on the green plate in front of them. Patients will be asked to replicate this position for each test. The static balance test will require that the subjects stand as quiet as possible during 35 seconds in 4 different conditions in the following order: (i) eyes open and easy counting, (ii) eyes closed and easy counting, (iii) eyes closed and counting in multiples of seven, and (iv) eyes closed and counting backward from 500 in multiples of seven.

The force platform, scale, and person altimeter will be calibrated every fortnight or more frequent. Data will be extracted, checked for any abnormal discrepancies, and saved on a secure driver frequently (at least every fortnight).

ELIGIBILITY:
Inclusion Criteria:

* Low back pain for more than 14 days

Exclusion Criteria:

* Signs of serious pathology (e.g. signs of fracture, cauda equina syndrome, malignancy, osteoporosis, or spinal inflammatory arthritis)
* Blindness
* Dyslexia and not able to reply questionnaires unassisted
* Pregnancy
* Not able to walk unassisted

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2017-02-04 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Medial-Lateral body sway | This is a cross sectional study all data will be collected during a 30 minute-session. The two balance tests for the primary outcome will be performed with a 1 minute interval.
  Additional medial-lateral body sway accessed by analysis of the Center of Pressure (CoP) position. Measured as the difference in medial-lateral CoP range (cm) between a difficult 30 sec. test (eyes closed and difficult counting backwards in multiples of seven) and an easy 30 sec. test (open eyes and easy counting forwards).

SECONDARY OUTCOMES:
Medial-Lateral body sway | This is a cross sectional study all data will be collected during a 30 minute-session. The three balance tests will be performed consecutively within 2 minutes interval.
  Additional medial-lateral body sway accessed by analysis of the Center of Pressure (CoP) position. Measured as the difference in medial-lateral CoP range (cm) between a medium 30 sec. test (eyes closed and counting forwards in multiples of seven), a medium-easy 30 sec. test (eyes closed and easy counting backwards), and an easy 30 sec. test (open eyes and easy counting forwards).
Medial-Lateral body sway | This is a cross sectional study all data will be collected during a 30 minute-session. The four balance tests will be consecutively within 3 minutes interval.
  Additional medial-lateral body sway will be accessed by analysis of the difference in CoP; velocity (cm/s) between a difficult 30 sec. test (eyes closed and difficult counting backwards in multiples of seven), a medium 30 sec. test (eyes closed and counting forwards in multiples of seven), a medium-easy 30 sec. test (eyes closed and easy counting backwards), and an easy 30 sec. test (open eyes and easy counting forwards).
Anterior-Posterior body sway | This is a cross sectional study all data will be collected during a 30 minute-session. The four balance tests will be consecutively within 3 minutes interval.
  Additional anterior-posterior body sway will be accessed by analysis of the difference in CoP; range (cm) between a difficult 30 sec. test (eyes closed and difficult counting backwards in multiples of seven), a medium 30 sec. test (eyes closed and counting forwards in multiples of seven), a medium-easy 30 sec. test (eyes closed and easy counting backwards), and an easy 30 sec. test (open eyes and easy counting forwards).
Anterior-Posterior body sway | This is a cross sectional study all data will be collected during a 30 minute-session. The four balance tests will be consecutively within 3 minutes interval.
  Additional anterior-posterior body sway will be accessed by analysis of the difference in CoP; velocity (cm/s) between a difficult 30 sec. test (eyes closed and difficult counting backwards in multiples of seven), a medium 30 sec. test (eyes closed and counting forwards in multiples of seven), a medium-easy 30 sec. test (eyes closed and easy counting backwards), and an easy 30 sec. test (open eyes and easy counting forwards).
Body sway area | This is a cross sectional study all data will be collected during a 30 minute-session. The four balance tests will be consecutively within 3 minutes interval.
  Additional sway area accessed by area of an ellipse fitted to the 95% confidence interval of the Center of Pressure position (cm2). Measured as the difference in area (cm2) between a difficult 30 sec. test (eyes closed and difficult counting backwards in multiples of seven), a medium 30 sec. test (eyes closed and counting forwards in multiples of seven), a medium-easy 30 sec. test (eyes closed and easy counting backwards), and an easy 30 sec. test (open eyes and easy counting forwards).

CONTACTS AND LOCATIONS:
Overall Officials: Allan Riis, PhD, Principal Investigator — Research unit for General Practice in Aalborg, Denmark
Locations (1):
- Sofiendal fysioterapi og kiropraktik, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No
The data analysed will be available from the corresponding author on reasonable request.

REFERENCES:
- [Background] Hoy D, March L, Brooks P, Blyth F, Woolf A, Bain C, Williams G, Smith E, Vos T, Barendregt J, Murray C, Burstein R, Buchbinder R. The global burden of low back pain: estimates from the Global Burden of Disease 2010 study. Ann Rheum Dis. 2014 Jun;73(6):968-74. doi: 10.1136/annrheumdis-2013-204428. Epub 2014 Mar 24. PMID 24665116
- [Background] Main CJ, Sowden G, Hill JC, Watson PJ, Hay EM. Integrating physical and psychological approaches to treatment in low back pain: the development and content of the STarT Back trial's 'high-risk' intervention (StarT Back; ISRCTN 37113406). Physiotherapy. 2012 Jun;98(2):110-6. doi: 10.1016/j.physio.2011.03.003. Epub 2011 Jun 12. PMID 22507360
- [Background] Sowden G, Hill JC, Konstantinou K, Khanna M, Main CJ, Salmon P, Somerville S, Wathall S, Foster NE; IMPaCT Back study team. Targeted treatment in primary care for low back pain: the treatment system and clinical training programmes used in the IMPaCT Back study (ISRCTN 55174281). Fam Pract. 2012 Feb;29(1):50-62. doi: 10.1093/fampra/cmr037. Epub 2011 Jun 27. PMID 21708984
- [Background] Hill JC, Whitehurst DG, Lewis M, Bryan S, Dunn KM, Foster NE, Konstantinou K, Main CJ, Mason E, Somerville S, Sowden G, Vohora K, Hay EM. Comparison of stratified primary care management for low back pain with current best practice (STarT Back): a randomised controlled trial. Lancet. 2011 Oct 29;378(9802):1560-71. doi: 10.1016/S0140-6736(11)60937-9. Epub 2011 Sep 28. PMID 21963002
- [Background] Foster NE, Mullis R, Hill JC, Lewis M, Whitehurst DG, Doyle C, Konstantinou K, Main C, Somerville S, Sowden G, Wathall S, Young J, Hay EM; IMPaCT Back Study team. Effect of stratified care for low back pain in family practice (IMPaCT Back): a prospective population-based sequential comparison. Ann Fam Med. 2014 Mar-Apr;12(2):102-11. doi: 10.1370/afm.1625. PMID 24615305
- [Background] Mientjes MI, Frank JS. Balance in chronic low back pain patients compared to healthy people under various conditions in upright standing. Clin Biomech (Bristol). 1999 Dec;14(10):710-6. doi: 10.1016/s0268-0033(99)00025-x. PMID 10545625
- [Background] Mok NW, Brauer SG, Hodges PW. Hip strategy for balance control in quiet standing is reduced in people with low back pain. Spine (Phila Pa 1976). 2004 Mar 15;29(6):E107-12. doi: 10.1097/01.brs.0000115134.97854.c9. PMID 15014284
- [Background] Salavati M, Mazaheri M, Negahban H, Ebrahimi I, Jafari AH, Kazemnejad A, Parnianpour M. Effect of dual-tasking on postural control in subjects with nonspecific low back pain. Spine (Phila Pa 1976). 2009 Jun 1;34(13):1415-21. doi: 10.1097/BRS.0b013e3181a3a917. PMID 19478663
- [Background] Maribo T, Schiottz-Christensen B, Jensen LD, Andersen NT, Stengaard-Pedersen K. Postural balance in low back pain patients: criterion-related validity of centre of pressure assessed on a portable force platform. Eur Spine J. 2012 Mar;21(3):425-31. doi: 10.1007/s00586-011-1981-5. Epub 2011 Aug 24. PMID 21863458